CLINICAL TRIAL: NCT03801304
Title: Open Label Phase II Trial to Evaluate Safety and Efficacy of Vinorelbine With Metronomic Administration in Combination With Atezolizumab as Second-line Treatment for Patients With Stage IV Non-small Cell Lung Cancer
Brief Title: Trial to Evaluate Safety and Efficacy of Vinorelbine With Metronomic Administration in Combination With Atezolizumab as Second-line Treatment for Patients With Stage IV Non-small Cell Lung Cancer
Acronym: VinMetAtezo
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: University Hospital, Brest (Other)
Collaborators: Groupe Francais De Pneumo-Cancerologie (Other); Roche Farma, S.A (Industry); Pierre Fabre Medicament (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: 29BRC18-0005 (VinMetAtezo)
Record Dates: First submitted 2019-01-07; First posted 2019-01-11 (Actual); Last update posted 2022-05-12 (Actual); Status verified 2022-05

CONDITIONS: Non-small Cell Lung Cancer
Keywords: immunotherapy; second line of chemotherapy
MeSH Terms: conditions — Carcinoma, Non-Small-Cell Lung | interventions — atezolizumab; Vinorelbine

STUDY DESIGN:
Intervention Model Description: * Atezolizumab will be administered of 1200 mg on day 1 of each 21-day cycle with IV infusions .
  * Vinorelbine at the dose of 40 mg per days will be administered on days 1, 3 and 5 of each week of the 21-day cycle.
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- Atezolizumab associated with vinorelbine (Experimental): * Atezolizumab will be administered with IV infusions. The first one will be a 60-min IV infusion; the subsequent infusions will last 30 minutes when well-tolerated at the dose of 1200 mg on day 1 of each 21-day cycle.
  * Vinorelbine capsules are taken orally on days 1, 3 and 5 of each week of the 21-day cycle. Vinorelbine will be administered at the dose of 40 mg per day on days 1, 3 and 5 of each week of the 21-day cycle. In case of toxicity, the dose will be decreased to 30 mg.
  Interventions: Drug: Atezolizumab; Drug: Vinorelbine

INTERVENTIONS:
Drug: Atezolizumab — Atezolizumab in IV infusions
Drug: Vinorelbine — Vinorelbine capsules

SUMMARY:
The majority of patients diagnosed with advanced NSCLC are treated with platinum-doublet chemotherapy regimens, except those harboring specific oncogenic drivers such as epidermal growth-factor-receptor (EGFR) mutations or anaplastic lymphoma kinase (ALK) rearrangements. In the second-line setting, response rates remain low and median survival rarely exceeds 10 months.

Over the past few years, several checkpoint inhibitors targeting programmed cell death protein-1 (PD1) or its ligand (PDL1) used as second-line therapies generated evidence of improving survival and, more recently, as first-line NSCLC treatment.

Although pembrolizumab (anti-PD1) was recently approved as first-line treatment for patients with at least 50% of their NSCLC cells expressing PDL1, many patients are still not benefiting from this first-line agent.

For patients with relapsed NSCLC, atezolizumab (anti-PDL1) prolonged survival compared to docetaxel in the phase II POPLAR and phase III OAK trials. Novel concepts of synergic action between immunotherapy and chemotherapy have emerged recently. However, those types of treatments are given for different durations: chemotherapy is allowed for only a short period (rarely exceeding 6 cycles), while anti-PDL1 can be continued for several months until loss of its clinical benefit.

Metronomic chemotherapy is defined as low-dose and frequent chemotherapy administration, without prolonged drug-free breaks. Metronomic administration of oral vinorelbine has been tested against breast cancer and advanced refractory NSCLC. The combination could have immunostimulatory effects: induction of immunogenic cancer-cell death, enhancement of antigen presentation through dendritic cell modulation, increased cancer-cell immunogenicity, preferential depletion of regulatory T cells, modulation of myeloid-derived suppressor cells, enhancement of the cytotoxic activity of immune-effector cells.

ELIGIBILITY:
Inclusion Criteria:

* Histologically confirmed NSCLC;
* Locally advanced and/or metastatic stage IV NSCLC (according to American Joint Committee on Cancers) or recurrent NSCLC);
* Patients without activating EGFR mutation or ALK rearrangement and ROS1 fusions.
* Subject has provided a formalin-fixed tumor-tissue sample of a tumor-lesion biopsy, either at the time of or after metastatic disease was diagnosed AND from a site not previously irradiated to assess for PDL1 status. Archived tissue may be acceptable or PDL1 status known;
* Progressive disease after first-line platinum-doublet-based chemotherapy according to RECIST V.1.1 with measurable lesion (RECIST V1.1);
* Age ≥18 years, either sex;
* Eastern Collaborative Oncology Group Performance status (ECOG PS) 0, 1 or 2;
* Life expectancy exceeds 12 weeks;
* No history of other malignancy within the last 5 years, except for adequately treated carcinoma in situ of the cervix or basal cell or spinocellular carcinoma of the skin;
* Adequate organ function, demonstrated by the following laboratory results within 3 weeks prior to teatment: Normal hepatic function: bilirubin <1.5 × normal (N), Alanine aminotransferase and Aspartate aminotransferase <2.5 × N or <5 × N if liver metastasis is present;
* Normal renal function (calculated creatinine clearance ≥45 mL/min);
* Normal calcemia;
* Normal hematological function (polynuclear neutrophils >1.5 G/L, platelets >100 G/L and hemoglobin>8g/dl);
* Women of child-bearing potential must use effective contraception;
* Men might be surgically sterile or accept to use an effective contraceptive procedure during and until 6 months after the treatment;
* Written informed consent to participate in the study
* Patient with social insurance

Exclusion Criteria:

* ECOG PS >2;
* Known hypersensitivity to immunotherapy;
* Small-cell lung cancer, bronchioloalveolar cancer, neuroendocrine cancer;
* Tumor harbors EGFR-sensitizing (activating) mutations or ALK translocations or ROS1 fusions and that justify treatment with targeted therapy ;
* Chemotherapy, hormonotherapy, immunotherapy or tyrosine-kinase inhibitors within the past 4 weeks prior to treatment with the trial drug;
* Radiotherapy (except bone or brain) within the past 3 months prior to baseline imaging;
* Medical contraindication to oral vinorelbine;
* Persistence of clinical adverse events with a grade > 2 related to prior treatment;
* Active brain metastases (e.g. stable for <4 weeks, no adequate previous radiotherapy, symptomatic, requiring anticonvulsants or corticosteroids)
* Concurrent radiotherapy, except for palliative bone irradiation.
* Other concurrent severe illnesses (congestive heart failure, unstable angina, significant arrhythmia or myocardial infarction <12 months before study entry);
* Active or prior documented autoimmune or inflammatory disorders;
* Active B hepatitis, HIV infection …;
* Psychiatric or neurological disorders preventing the patient from understanding the nature of the trial;
* Grade-3 peripheral neuropathy;
* Uncontrolled infection;
* Interstitial lung disease or pneumonitis requiring steroid management;
* Corticosteroid therapy exceeding 10 mg/day;
* Other severe organic disorders not allowing inclusion in the trial;
* Malabsorption syndrome;
* Pregnancy or breast-feeding;
* Follow-up not possible; and incarcerated or institutionalized patients.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 80 (Actual)
Dates: Start 2019-01-24 (Actual); Primary Completion 2021-01-04 (Actual); Study Completion 2022-02-23 (Actual)

PRIMARY OUTCOMES:
Occurrence of death or progression of the disease | 4 months
  To evaluate the occurrence of death or progression of the disease

SECONDARY OUTCOMES:
Emergence of adverse events (Safety and tolerability) | 12 months
  To evaluate the safety outcomes, tolerability, adverse events frequency
Occurrence of death | 12 months
  To evaluate the occurrence of death over 12 months of follow-up
Objective Response Rate | 4 months
  To evaluate the objective Response Rate and Disease Control Rate
Following of the quality of life | 12 months
  The scale EuroQol 5 dimensions (EDQ5) is used to evaluate the quality of life. The EQ-5D scale is a standardised measure of health status to provide a simple, generic measure of health for clinical and economic appraisal, whih is divided by the EQ-5D descriptive system (mobility, self care, usual activities, pain/discomfort, anxiety/depression) and the EQ Visual Analogue scale (EQ VAS). Each dimension has 5 levels (no problems, slight problems, moderate problems, severe problems, and extreme problems).
Following of the quality of life | 12 months
  The EORTC QLQ-C30 is a questionnaire with 30 questions developed to assess the quality of life of cancer patients. An essential aspect of the "modular" approach to QOL assessment adopted by the EORTC Quality of Life Group is the development of modules specific to tumour site, treatment modality, or a QOL dimension, to be administered in addition to the core questionnaire (EORTC QLQ-C30).

CONTACTS AND LOCATIONS:
Locations (13):
- France (13):
  - CH Aix en Provence, Aix-en-Provence
  - CHRU de Brest - Hôpital Morvan, Brest
  - CLCC Caen, Caen
  - CH de Créteil, Créteil
  - Ch La Roche Sur Yon, La Roche-sur-Yon
  - CHU de Limoges - Hôpital DUPUYTREN, Limoges
  - CH MEAUX, Meaux
  - CH Pringy, Pringy
  - CH Quimper, Quimper
  - CHU de Rennes, Rennes
  - CHU Rouen, Rouen
  - CH Saint-Brieuc, Saint-Brieuc
  - Hia Saint Anne, Toulon

IPD SHARING:
Plan to Share IPD: Yes
All collected data that underlie results in a publication
Supporting Information: Study Protocol
Time Frame: Data will be available beginning three years and ending fifteen years following the final study report completion
Access Criteria: Data access requests will be reviewed by the internal committee of Brest UH. Requestors will be required to sign and complete a data access agreement.

REFERENCES:
- [Derived] Vergnenegre A, Monnet I, Bizieux A, Bernardi M, Chiapa AM, Lena H, Chouaid C, Robinet G. Open-label Phase II trial to evaluate safety and efficacy of second-line metronomic oral vinorelbine-atezolizumab combination for stage-IV non-small-cell lung cancer - VinMetAtezo trial, (GFPCdouble dagger 04-2017). Future Oncol. 2020 Feb;16(4):5-10. doi: 10.2217/fon-2019-0730. Epub 2020 Jan 2. PMID 31894704